CLINICAL TRIAL: NCT04240639
Title: A Study of MRI/US Fusion Imaging and Biopsy in Combination With Nanoparticle Directed Focal Therapy for Ablation of Prostate Tissue
Brief Title: An Extension Study MRI/US Fusion Imaging and Biopsy in Combination With Nanoparticle Directed Focal Therapy for Ablation of Prostate Tissue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanospectra Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-PC-002.1
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms of the Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AuroShell particle infusion (Experimental): Single intravenous infusion of AuroShell particles 12 to 36 hours prior to MRI/US guided laser irradiation using an FDA cleared laser and an interstitial optical fiber diffuser.
  Interventions: Device: AuroShell particle infusion

INTERVENTIONS:
Device: AuroShell particle infusion — Infuse AuroShell particles for irradiation by AuroLase laser to ablate neoplasms of the prostate.

SUMMARY:
To determine the efficacy of using MRI/US fusion imaging technology to direct focal ablation of prostate tissue using nanoparticle-directed laser irradiation.

DETAILED DESCRIPTION:
This is an open-label, multi-center, single-dose study of AuroLase Therapy in the focal ablation of prostate tissue via nanoparticle directed irradiation.

The patient population consists of men with low to intermediate risk localized prostate cancer with MRI visible and confirmed focal areas of prostate cancer using MR US Fusion Guided Biopsy.

There is one arm/group to this study: Up to sixty (60) patients will receive a single intravenous infusion of AuroShell particles 12 to 36 hours prior to MRI/US guided laser irradiation using an FDA cleared laser and an interstitial optical fiber diffuser.

Efficacy and acute volume of ablation will be assessed by contrast-enhanced MRI 48 - 96 hours after laser illumination to allow time for the appearance of coagulative necrosis and prior to reconfiguration of tissue by lytic action. An appearance of a 'void' (e.g., lack of contrast in ablation zone) on MRI would be more generally expected than lesion shrinkage.

Efficacy of focal ablation of prostate tissue will be assessed by MRI /Ultrasound guided target biopsy 6 months after laser treatment and at 1 year via MRI /Ultrasound guided target biopsy in combination with standard systematic biopsy. Per standard of care, patient follow up will continue beyond the one year study visit but will be outside the scope of the study. Patients will be consented for up to 5 years in order to track their disease status and progression or recurrence if any.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented histological or cytological evidence of tumor(s) of the prostate.
* Patients must be ≥ 45 years of age
* Patients or their legal representative must be able to read, understand and sign an informed consent
* Organ confined clinical T1C or clinical T2a prostate cancer that is visualized on MR imaging
* Prostate cancer is diagnosed by MR image guided biopsies
* Gleason Score ≤ 7; and 2 or less positive lesions on prior MR US fusion guided prostate biopsy.
* A non MRI visible cancer detected via systematic standard biopsy will not be considered an exclusion condition provided the non-MRI visible cancer is singularly located in the contralateral hemisphere of the prostate; is Gleason 6 cancer; and comprises no more than 6mm linear extent of cancer in a single core on standard biopsy.
* If any standard biopsy cores are positive on the same hemisphere of the prostate gland, they must be confirmed as likely to form a contiguous lesion with the target lesion detected on MRI and therefore be from the same location in the prostate as MR lesion was biopsied and proven to be cancerous. (e.g., Left/Right, Base, Mid Gland, Apex).
* Prior mpMRI results dated within 120 days prior to ablation.
* No metastatic disease as per NCCN guidelines (www.nccn.org) - Bone scan indicated to r/o metastatic disease if clinical T1 and PSA > 20 or T2 and PSA > 10
* PSA < 15 ng/ml or PSA density < 0.15 ng/ml2 in patients with a PSA > 15 ng/ml
* The patient has given written informed consent after the nature of the study and alternative treatment options have been explained.

Exclusion Criteria:

* Patients with known hypersensitivity to any of the components of the PEGylated AuroShell suspension (polyethylene glycol, gold).
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within a period of 5 half-lives of the investigational therapy in questions prior to the day of dosing with PEGylated AuroShell particles (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Patients with evidence of an active bacterial infection or with a fever ≥ 38.5 ºC (101.3 ºF) within 3 days of the first scheduled day of dosing
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* The presence of 3 or more MR Visible lesions positive on biopsy.
* The presence of extra capsular, seminal vesicle invasion or metastatic disease.
* Patient is unable to tolerate MRI (foreign body; i.e. pacemaker or other implanted device; claustrophobia; inability to tolerate rectal coil, etc.…)
* Patient with inability to follow up.
* History of prior treatment for prostate cancer.
* Acute urinary tract infection.
* Lower urinary tract symptoms defined by International Prostate symptom score (IPSS) > 20
* Patients with renal insufficiency with an estimated glomerular filtration (EGF) <= 30 are excluded, as they will not be able to undergo gadolinium enhance MRI.
* Patients with acute or chronic hepatic dysfunction as evidenced by clinically important (> grade 1) changes in AST, ALT, bilirubin, or albumin, or either ALP or GGT values.
* Patients with uncontrolled coagulopathies who are at increased risk of bleeding, or with abnormal PT (INR) or PTT.
* Altered mental status preventing consent or answering questions during conduct of the trial will be excluded for safety purposes.
* Other medical or surgical conditions, especially involving the cardiac, respiratory, renal or hepatic organ systems that would either be unsafe for the patient, would limit study participation, or that would impede the determination of causality of any adverse events experienced during the conduct of this study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Evidence of efficacy of focal ablation of clinically significant targeted prostate lesion(s) confirmed using 3T MRI/Ultrasound guided biopsy 3 months after treatment. | Six Months
  To determine the efficacy at 6 months post treatment of using MRI/US fusion imaging technology to direct focal ablation of prostate tissue using nanoparticle-directed laser irradiation. MRI/US Fusion biopsy of the treatment zone at both time points post treatment will assess presence of clinically significant prostate disease as confirmed by pathology.
Evidence of efficacy of focal ablation of clinically significant targeted prostate lesion(s) | One Year
  To determine the efficacy at 1-year post treatment of using MRI/US fusion imaging technology to direct focal ablation of prostate tissue using nanoparticle-directed laser irradiation. MRI/US Fusion biopsy of the treatment zone at both time points post treatment will assess presence of clinically significant prostate disease as confirmed by pathology.

SECONDARY OUTCOMES:
Adverse Events | Day One to One Year
  Any adverse device effects attributable to near infrared illumination of the prostate following AuroShell particle infusion.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Urology, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Lenox Hill/Northwell Health System, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Medical School at Houston, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided